CLINICAL TRIAL: NCT04617977
Title: Interdependent Quality of Life in Parent-Child Dyads Adjusting to Eczema: Effects of a Randomized Controlled Trial of the Integrative Body-Mind-Spirit Group Intervention
Brief Title: Integrative Body-Mind-Spirit Intervention for Families With Children Suffering From Eczema
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Celia Hoi-Yan Chan, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA2001001
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Eczema; Dermatitis, Atopic
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parent-child I-BMS intervention group (Experimental): Children with eczema and their parent caregivers will attend the six sessions simultaneously in a parallel group format. Parent caregivers will attend the parents group in the first 2.5 hours; while children will attend the children group in the first 2.5 hours. Both parents and children will later reunite in the joint group in the final 0.5 hours.
  Interventions: Behavioral: I-BMS for families with children suffering from eczema
- Parent only I-BMS intervention group (Experimental): Only parent caregivers of children with eczema will attend the six sessions. The content of the 2.5-hour parents group will be the same as the one in Arm 1 (Parent-child I-BMS intervention group), with an additional 0.5 hour of reflective discussion among group members. The children group will simultaneously attend a group activity class in a separate room for 3 hours.
  Interventions: Behavioral: I-BMS for families with children suffering from eczema
- Parent only health education active control group (Active Comparator): Only parent caregivers of children with eczema will attend the six sessions. Each session consists of teaching in the first 2.5 hours and Q&A in the final 0.5 hour. The children group will simultaneously attend a group activity class in a separate room for 3 hours.
  Interventions: Behavioral: Health education for parents whose children have eczema

INTERVENTIONS:
Behavioral: I-BMS for families with children suffering from eczema — It is a strength-based, family system approach to aid empowerment of individuals. It focuses on the interplay between physical and emotional well-being, the spiritual transformation of adverse life experiences, and the acceptance of adversity through reflection on the philosophical concepts of forgiveness and letting go. It integrates Western therapeutic techniques and Eastern philosophies to develop spiritual transformation through suffering and pain under a meaning-oriented framework. It consists of six three-hour consecutive weekly sessions: (1) awareness of body-mind connection; (2) regulation of emotion; (3) acknowledgement of the gains and losses in the caregiving or illness experience; (4) appreciation of self and others; (5) cultivation of acceptance; and (6) meaning reconstruction of caregiving or illness experience.
  Arms: Parent only I-BMS intervention group; Parent-child I-BMS intervention group
Behavioral: Health education for parents whose children have eczema — It focuses on practical eczema management. It serves as a control for group effect between conditions. It consists of six three-hour sessions: (1) information about the physiology of eczema and its health impact; (2) recognition and avoidance of trigger factors and daily skin care; (3) dealing with itching and scratching; (4) stage-related treatment of symptoms and unconventional therapies; (5) general child nutrition, food allergies in eczema, and different forms of diets; and (6) self-management plan and problems in integrating into daily routine.
  Arms: Parent only health education active control group

SUMMARY:
This randomized controlled trial aims to examine the efficacy of two integrative body-mind-spirit interventions, compared to a health education active control, in promoting adaptive emotional regulation and quality of life of children with eczema and their parent caregivers in Hong Kong. It also aims to examine the interdependent associations between children and their parent caregivers' baseline primary outcomes and the post-intervention changes in primary outcomes.

DETAILED DESCRIPTION:
Childhood eczema is a significant pediatric health crisis in Hong Kong. It not only has adverse psychosocial impacts on children, but also poses tremendous burden for their parent caregivers. The interdependence of family members calls for a systemic family-based psychosocial intervention.

An integrative body-mind-spirit (I-BMS) intervention for families with children suffering from eczema has been developed, and its initial results are promising. Compared to the waitlist control group, parent caregivers in the I-BSM intervention group reported significantly more improvements in perceived stress, depression and well-being. Likewise, children in the I-BSM intervention group reported significantly more improvements in somatic eczema severity, generalized anxiety, social phobia and emotional regulation. It is not clear, however, if the I-BMS intervention delivered only to the parent caregivers would be: (1) as efficacious as the I-BMS intervention delivered to both the parent caregivers and children, and (2) more efficacious than the health education delivered only to the parent caregivers, in improving their emotional regulation and quality of life. This three-arm parallel randomized controlled trial (RCT) aims to examine the efficacy of two I-BMS interventions (one delivered to both parents and children, one delivered to parents only), compared to a health education active control (delivered to parents only), in promoting adaptive emotional regulation and quality of life of children with eczema and their parent caregivers. This RCT also aims to examine the interdependent associations between children and their parent caregivers' baseline primary outcomes and the post-intervention changes in primary outcomes.

One hundred and ninety-two parent-child dyads will be recruited through hospitals and non-governmental organizations in various districts in Hong Kong. Each dyad will complete an individual pre-group screening interview. Those who meet the eligibility criteria will be randomized in a ratio of 1:1:1 into one of the three arms, hence, each arm will have 64 parent-child dyads. Arm 1 is I-BMS intervention delivered to both children and their parent caregivers. Arm 2 is I-BMS intervention delivered to parent caregivers only. Arm 3 is health education delivered to parent caregivers only. Each arm consists of six weekly three-hour sessions. A computer-generated list of random numbers will be used to perform randomization. The primary outcomes are changes over the measurement points in quality of life and emotional regulation. The secondary outcomes include changes over the measurement points in depression, anxiety, stress, parent-child relationship, holistic well-being, caregiver burden, and perceived eczema severity. Assessments will be administered at baseline, post-intervention, and 6-week follow up. Important adverse events, if any, will be documented. Mixed factorial ANCOVAs based on intention-to-treat principle will be conducted to examine the efficacy of the two I-BMS interventions.

Seven hypotheses are generated. First, it is hypothesized that, after the intervention, participants in the two I-BMS intervention groups will report significantly more improvements in emotional regulation and quality of life than those in the health education active control group. Second, it is hypothesized that there is no significant difference between the two I-BMS intervention groups in terms of post-intervention improvements in emotional regulation and quality of life. Third, it is hypothesized that the post-intervention improvements in emotional regulation and quality of life will be maintained at 6-week follow-up for the two I-BMS intervention groups, but not for the health education active control group. Fourth, it is hypothesized that children's baseline quality of life is predicted by their own baseline emotional regulation and by their parents' baseline quality of life. Fifth, it is hypothesized that parents' baseline quality of life is predicted by their own baseline emotional regulation and by their children's baseline quality of life. Sixth, it is hypothesized that children's post-intervention improvements in quality of life are predicted by their own post-intervention improvements in emotional regulation and their parents' post-intervention improvements in quality of life. Seventh, it is hypothesized that parents' post-intervention improvements in quality of life are predicted by their own post-intervention improvements in emotional regulation and their children's post-intervention improvements in quality of life.

ELIGIBILITY:
Inclusion Criteria (Children):

* age 6-12
* are diagnosed with atopic dermatitis as assessed by the doctors (ICD-10 Revision codes L20-L30)
* are able to communicate in Cantonese
* give their consent to participate in this RCT
* obtain parental consent to participate in this RCT

Inclusion Criteria (Parent caregivers):

* are the primary caregivers of the child participants
* are able to communicate in Cantonese
* give their consent to participate in this RCT

Exclusion Criteria (Children):

- are diagnosed with Autism Spectrum Disorder or Attention Deficit Hyperactivity Disorder

Exclusion Criteria (Parent caregivers):

* exhibit a history of family abuse
* present with clinically significant psychiatric morbidity such as psychosis

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes over the measurement points in the Family Dermatology Life Quality Index | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 10 items. It measures how much a child with atopic dermatitis affects the quality of life of their parent caregivers. Scores range from 0 to 30, where a high score represents a greater effect on the life of the parent caregiver.
Changes over the measurement points in the Children's Dermatology Life Quality Index | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 10 items. It measures the impact of atopic dermatitis on the lives of children. Scores range from 0 to 30, where a higher score represents a greater impact on the child's life.
Changes over the measurement points in the Cognitive Emotion Regulation Questionnaire - Short Version | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 18 items. It measures the specific cognitive emotion regulation strategies parent caregivers have used when caring for their children. It has nine subscales, namely, self-blame, other-blame, rumination, catastrophizing, putting into perspective, positive refocusing, positive appraisal, acceptance and planning. Subscale scores range from 2 to 10, where a higher score represents more usage of a specific cognitive emotion strategy.
Changes over the measurement points in the Short Version of the Cognitive Emotion Regulation Questionnaire for Spanish Kids | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 18 items. It measures the specific cognitive emotion regulation strategies children have used to cope with their illness experience. It has nine subscales, namely, self-blame, other-blame, rumination, catastrophizing, putting into perspective, positive refocusing, positive appraisal, acceptance and planning. Subscale scores range from 2 to 10, where a higher score represents more usage of a specific cognitive emotion strategy.

SECONDARY OUTCOMES:
Changes over the measurement points in the Hospital Anxiety and Depression Scale | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 14 items. It measures parent caregivers' emotional states of depression and anxiety. It has two subscales, namely, depression and anxiety. Subscale scores range from 0 to 21, where a higher score represents a higher level of depression or anxiety.
Changes over the measurement points in the Revised Child Anxiety and Depression Scale - Short Version | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 25 items. It measures children's emotional states of depression and anxiety. The depression subscale has 10 items, its scores range from 0 to 30, where a higher score represents a higher level of depression. The anxiety subscale has 15 items, its scores range from 0 to 45, where a higher score represents a higher level of anxiety.
Changes over the measurement points in the Perceived Stress Scale for Children | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 14 items. It measures children's emotional states of stress. One item is for illustration purposes and is not scored. Scores range from 0 to 39, where a higher score represents a higher level of stress.
Changes over the measurement points in the Perceived Stress Scale | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 10 items. It measures parent caregivers' emotional states of stress. Scores range from 0 to 40, where a higher score represents a higher level of stress.
Changes over the measurement points in the Parent-Child Relationship Questionnaire - Personal Relationship Subscale (Parent Form) | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 10 items. It measures parent caregivers' perception of their relationship quality with their children. Scores range from 10 to 50, where a higher score represents a better parent-child relationship.
Changes over the measurement points in the Parent-Child Relationship Questionnaire - Personal Relationship Subscale (Child Form) | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 10 items. It measures children's perception of their relationship quality with their parent caregivers. Scores range from 10 to 50, where a higher score represents a better parent-child relationship.
Patient-Oriented Eczema Measure for Child (Parent Form) | Baseline, post-intervention: 6 weeks after intervention initiation, 6-week follow up
  It has 7 items. It measures parent caregivers' perception of their children's eczema severity. Scores range from 0 to 28, where a higher score represents more severe eczema.

OTHER OUTCOMES:
Satisfaction with Treatment Program Scale | Post-intervention: 6 weeks after intervention initiation
  It has 5 items. It measures parent caregivers' satisfaction with the intervention. Scores range from 5 to 25, where a higher score represents lower satisfaction.
Demographics | Baseline
  Single items will be used to measure children's demographics (age, gender, and education level), as well as their parent caregivers' demographics (age, gender, education level, marital status, employment status, household income, type of housing, number of children).
Childhood eczema onset age | Baseline
  One single item will be used to measure the onset age of childhood eczema.
Current treatment for childhood eczema | Baseline
  Seven items will be used to measure the types of eczema treatments the children are receiving.
Cross-condition contamination check | Post-intervention: 6 weeks after intervention initiation
  Two items will be used to control for the confounding effect of unexpected exposure to I-BMS intervention materials during the trial on primary outcomes. Only participants in the health education active control group (arm 3) will complete it.
Presence of other clinical co-morbidities | Baseline
  Two items will be used to gather information about the presence of other clinical co-morbidities (e.g., allergy) among the children

CONTACTS AND LOCATIONS:
Overall Officials: Celia Hoi-Yan Chan, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Social Work and Social Administration, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hui VKY, Chan CHY, Fung YL, Chan CLW, Luk MSK. Efficacy of the integrative Body-Mind-Spirit group intervention for improving quality of life in parent-child dyads adjusting to atopic dermatitis: protocol for a randomised controlled trial. BMJ Open. 2022 Mar 16;12(3):e059150. doi: 10.1136/bmjopen-2021-059150. PMID 35296490